CLINICAL TRIAL: NCT00279227
Title: Role of Epicardial Adipose Tissue in Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Organization: McMaster University (Other)
Other Study IDs: EPICARD Study
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-01

CONDITIONS: Coronary Artery Disease; Obesity
Keywords: coronary artery disease; epicardial adipose tissue; epicardial fat; obesity
MeSH Terms: conditions — Coronary Artery Disease; Obesity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
We sight to evaluate whether patients with coronary artery disease (CAD) have more epicardial fat than patients without CAD, which would suggest that epicardial fat may be more than an "innocent bystander" and be actively involved in the disease process. Its role as a modulator of vascular response and myocardial function could potentially lead to new areas of cardiac research. We also sight to evaluate whether epicardial fat from patients with CAD releases more adipokines than subcutaneous fat from these patients which could prompt studies into the differential regulation of adipokine secretion in this tissue. Thus for e.g., the use of thiazolidinediones (glitazones), statins, ARBs or other compounds that can specifically modulate adipokine secretion could be explored to determine their benefit in ameliorating the effects attributable to increased epicardial fat.

ELIGIBILITY:
Inclusion Criteria:

* All patients elegible for elective cardiac surgery are elegible
* Ability to provide written informed consent in accordance with GCP guidelines and local legislations.
* > 18 years of age

Exclusion Criteria:

* Control patients will not have clinical signs of CAD and will show normal coronary arteries on angiography.
* Any medical, social or geographic condition, which, in the opinion of the investigator would not allow safe or reliable completion of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Arya M Sharma, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - Cardiovascular Obesity Research and Management Center, Hamilton, Ontario, Canada